CLINICAL TRIAL: NCT06534047
Title: Integrating Transcranial Magnetic Stimulation as a Treatment for Nicotine Dependence in the Clinic: A Pragmatic, Hybrid Effectiveness-Implementation Trial
Brief Title: Transcranial Magnetic Stimulation for Nicotine Dependence: An Effectiveness-Implementation Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-018
Record Dates: First submitted 2024-06-07; First posted 2024-08-02 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2024-12

CONDITIONS: Tobacco Use Disorder; Psychiatric Disorder; Nicotine Dependence
Keywords: Repetitive Transcranial Magnetic Stimulation; Nicotine Dependence; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Mental Disorders; Smoking Cessation | interventions — Transcranial Magnetic Stimulation; Nicotine Replacement Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Hybrid type 1 Implementation effectiveness trial. Open label, randomized, parallel group
Masking Description: This is an open-label trial, so there will be no blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Repetitive Transcranial Magnetic Stimulation (rTMS) Intervention (Experimental): Treatment course consisting of daily treatment, 5 days per week, for 3 weeks, followed by once weekly treatments for 3 weeks, for a total of 18 treatment sessions over 6 weeks.
  Interventions: Device: Brainsway H4 deep Repetitive Transcranial Magnetic Stimulation (rTMS) coil
- Treatment as Usual (Active Comparator): Treatment with Nicotine Replacement Therapy (NRT) and/or adjunctive counselling will be provided by their clinical team through the Smoking Treatment for Ontario Patients (STOP) Program. All treatments will be delivered by study physicians in the Nicotine Dependence Clinic at CAMH, all of whom administer NRT through the STOP program.
  Interventions: Drug: Nicotine replacement

INTERVENTIONS:
Device: Brainsway H4 deep Repetitive Transcranial Magnetic Stimulation (rTMS) coil — An rTMS treatment course consisting of daily treatment, 5 days per week, for 3 weeks, followed by once weekly treatments for 3 weeks, for a total of 18 treatment sessions over 6 weeks.
  Sixty trains of 30 pulses each (total 1,800 pulses) will be applied at 10 Hz, for 3 second trains, with a 15 second inter-train interval, for approximately 18 minutes of treatment time.
  At each rTMS treatment session, prior to stimulation, participants will undergo a smoking craving provocation procedure where they will be asked to close their eyes and imagine one of their triggers for 30 seconds. Following this they will watch a presentation of smoking pictures for 2 minutes and 30 seconds. Thus, the entire craving provocation procedure will be 3 minutes prior to stimulation start.
  Brief behavioural support will be available to the participant on a weekly basis by a trained research staff member.
  Other Names: Deep TMS
  Arms: Repetitive Transcranial Magnetic Stimulation (rTMS) Intervention
Drug: Nicotine replacement — Each participant will receive individualized NRT treatment through the advice of their study physician for 6 weeks. The study physician, in discussion with the participant, will decide the type, dosage, and combination of NRT to provide to the participant.
  NRT provided can include:
  * Patch (7mg, 14mg, and 21mg)
  * Gum (2mg)
  * Lozenge (2mg)
  * Inhaler (10mg; 4mg of nicotine delivered)
  Other Names: Treatment As Usual
  Arms: Treatment as Usual

SUMMARY:
Tobacco smoking is the leading preventable cause of morbidity and mortality worldwide. However, currently available treatments, including standard pharmacotherapy and behavioural support, are limited in their efficacy, tolerability, and acceptability by patients. Additionally, tobacco use is substantially higher in individuals with comorbid mental illness, constituting a particularly vulnerable population. As such, the development of multiple evidence-based treatments for smoking cessation is of upmost importance.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain-based approach in which alternating magnetic fields are applied to the scalp to induce electrical currents in cortical tissue. As it can modulate neural circuits implicated in neuropsychiatric disorders, it is a promising brain-based approach in the treatment of substance use disorders. Recently, a deep TMS coil has been cleared by the Food and Drug Administration (FDA) as efficacious for tobacco use disorder, representing the first rTMS indication for addictions. Before adoption of this intervention into smoking cessation clinics, it is important to investigate whether implementation of rTMS into clinical care is feasible, acceptable, and appropriate for patients receiving care for nicotine dependence.

The objective of this study is to compare the effectiveness of rTMS versus treatment as usual for patients with psychiatric disorders seeking treatment for smoking cessation. Also, barriers to the implementation of rTMS in routine clinical care will be examined by speaking with patients and health care providers on their experience with rTMS.

DETAILED DESCRIPTION:
The objective is to pilot a pragmatic, randomized, comparative effectiveness trial of rTMS, compared to treatment as usual (TAU), for smoking cessation in individuals with psychiatric comorbidities, using a type 1 hybrid effectiveness-implementation design. Participants will be included if they meet DSM-5 criteria for mood disorders, anxiety disorders, psychotic disorders, posttraumatic stress disorder, obsessive compulsive disorders, or other substance use disorders. Those that undergo rTMS treatment will be offered open-label rTMS treatment with the FDA and Health Canada approved Brainsway deep TMS (dTMS) coil which includes 3 weeks of daily on-site rTMS treatments followed by 3 weeks of weekly treatments. Those that undergo TAU will receive nicotine replacement therapy and counselling through the supervision of a study physician.

ELIGIBILITY:
Inclusion Criteria:

Patient Participants:

The patient participant must meet all the inclusion criteria to be eligible for this study:

1. Able to provide informed consent.
2. Age 18-70.
3. Self-reported daily tobacco cigarette consumption.
4. Meet DSM-5 criteria for a psychiatric disorder that includes one of the following: mood disorders (e.g. major depressive disorder, bipolar disorder), anxiety disorders (e.g. panic disorder, social anxiety disorder), psychotic disorders (e.g. schizophrenia), posttraumatic stress disorder, obsessive compulsive disorders, or other substance use disorders (e.g. alcohol use disorder) as determined by the Structured Clinical Interview for DSM-5 Disorders, Research Version (SCID-5 RV).
5. Interested in using either Repetitive Transcranial Magnetic Stimulation (rTMS) or nicotine replacement therapy as a smoking cessation treatment.
6. Intending on quitting smoking within the next 30 days.

Exclusion Criteria:

Patient Participants:

1. Contraindication to rTMS according to the TMS Adult Safety Screen (TASS) and PI review.
2. Have any intracranial implant (e.g., aneurysm clips) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
3. Pregnant or intending to be pregnant during the study.
4. A history of a primary seizure disorder, seizure associated with an intracranial lesion, recurrent seizures related to substance intoxication or withdrawal or recent seizure within the last 6 months.
5. Space occupying intracranial lesion.
6. Any generalized skin disorders precluding the use of the nicotine patch.
7. Any known hypersensitivity or allergies to the nicotine patch.
8. Any known life-threatening arrhythmias or severe/worsening angina pectoris.
9. Within two weeks of experiencing a myocardial infarction or cerebral vascular accident.
10. Currently using or has used nicotine replacement therapy within the past two weeks.
11. Diagnosed with a terminal illness
12. Current regular use of e-cigarettes or other vaping devices containing nicotine and not willing to stop using these devices for the duration of the study.
13. Acutely unstable medical, psychiatric, or substance use disorder comorbidity with safety concerns at the discretion of the PI or study physician.
14. Previous treatment with rTMS for smoking cessation
15. Treatment with nicotine replacement therapy anytime within the last 1 month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of conducting a pragmatic, hybrid effectiveness implementation trial of Repetitive Transcranial Magnetic Stimulation (rTMS) versus treatment as usual (TAU). | Through study completion, an average of 2 years
  Recruitment over the 2-year study period will be measured, with a target sample of 40. Retention will be determined by the proportion of people who complete 50% of the treatments.

SECONDARY OUTCOMES:
Estimate the difference in effectiveness between Repetitive Transcranial Magnetic Stimulation (rTMS) and Treatment As Usual (TAU) on smoking cessation rates in real world patients with psychiatric comorbidities. | After completion of the intervention (rTMS or TAU; up to 6 weeks)
  Self-reported 4-week continuous quit rate and long follow-up continuous quit rate (biochemically verified by urine nicotine/tobacco metabolite collection and analysis at end of treatment and the long follow-up).
Estimate the implementation of Repetitive Transcranial Magnetic Stimulation (rTMS) in routine clinical care. | Through study completion, an average of 2 years
  Semi-structured interviews with NDC patients and healthcare providers to better understand the collaborative nature and necessary communication components involved in shared treatment decision-making for rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Victor M Tang, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada